CLINICAL TRIAL: NCT07150442
Title: The Effects of Platelet Rich Plasma Adjuvant to Type I/III Collagen Ratio, Matrix Metalloproteinase-2 and Matrix Metalloproteinase-9 in Pelvic Organ Prolapse Repair
Acronym: POP PRP MMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andalas University (Other)
Collaborators: Faculty of Medicine, Andalas University (Unknown); Dr. M Djamil Hospital, Padang (Unknown)
Responsible Party: Principal Investigator, Yulia Margaretta Sari, MD, Andalas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DP.04.03/D.XIV.10.1/301/2025; DP.04.03/D.XIV.10.1/301/2025 (Other: Health Research Ethic Committee M Djamil Hospital Padang Indonesia)
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Pelvic Organ Prolapse Vaginal Surgery; Platelet Rich Plasma Injection
Keywords: Pelvic organ prolapse surgery; Platelet rich plasma injection; Type I/III collagen ratio; MMP-2; MMP-9; Randomized controlled trial

STUDY DESIGN:
Intervention Model Description: Two group will receive different intervention One group will receive pelvic organ prolapse surgery and Platelet Rich Plasma injection One group will receive pelvic organ prolapse surgery and Placebo injection
Who Masked: Participant
Masking Description: Only participants are masked in this study. Care provider can not be blind because the operator it self inject PRP , meanwhile PRP have different colour to placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): patient who receive POP surgery and PRP injection
  Interventions: Procedure: POP surgery and PRP injection
- Group B (Experimental): patient who receive POP surgery and placebo injection
  Interventions: Procedure: POP surgery and placebo injection

INTERVENTIONS:
Procedure: POP surgery and PRP injection — Patient who undergo POP surgery will receive PRP injection
  Arms: Group A
Procedure: POP surgery and placebo injection — patient who receive POP surgery and placebo injection
  Arms: Group B

SUMMARY:
The goal of this clinical trial is to analyze the effect of Platelet Rich Plasma (PRP) Adjuvant To Type I/III Colagen Ratio, MMP-2 and MMP-9 in Pelvic Organ Prolapse Repair.

The main questions it aims to answer are:

Does the PRP Adjuvant affect type I/III Colagen Ratio, MMP-2 and MMP-9 in Pelvic Organ Prolapse Repair? Researchers will compare patient who undergo prolapse surgery with PRP adjuvant versus patient who undergo prolapse surgery without PRP adjuvant (placeebo)

Participants will:

Patient will undergo pelvic organ prolapse reconstrucion surgery and punch biopsy and injection of PRP will perform in anterior vaginal mucosa at Pubocervical area. The second biopsy will attempt in 8 weeks post operative. imunohistochemistry examination will be done to compare the type I/III Colagen Ratio, MMP-2 and MMP-9 before and after surgery.

DETAILED DESCRIPTION:
1. Prepare tools and materials for the research.
2. Align perceptions with the research team to conduct well-guided interviews.
3. Patients who meet the inclusion and exclusion criteria will be given an explanation and a research information sheet and asked for consent to participate in the study.
4. Subjects who agree to participate in the study will then undergo a urogynecological medical record and gynecological physical examination, pelvic floor muscle strength, and POP Q.
5. Randomization of study subjects will be performed.
6. Participants are unaware of whether they would receive PRP therapy or a placebo.
7. The study subjects were hospitalized in preparation for surgery, in accordance with the regulations of the hospital where the study subjects were located.
8. PRP was prepared from the patient's own blood on the day of surgery. Blood was drawn no later than one hour before surgery. Twenty milliliters of blood was collected for processing into PRP.
9. Participant undergo pelvic organ prolapse surgery as a medically indicated treatment for pelvic organ prolapse.
10. Punch biopsies were performed on the anterior vaginal mucosa located in the Fascia Pubocervicalis area, 6 mm deep. The tissue was sent in a special medium to the Anatomical Pathology Laboratory of Dr. M. Djamil General Hospital.
11. PRP or placebo injections were administered based on a random number sequence determined by block randomization among subjects undergoing POP surgery in the Surgical Unit of the hospital where the study subjects were located.
12. The PRP preparation was placed in a 5 cc syringe.
13. The placebo preparation, containing NaCl solution, was placed in a 5 cc syringe.
14. The injection was performed by the POP surgery operator into the anterior vaginal wall to a depth of approximately 1-1.5 cm, estimating the location of the Fascia Pubocervicalis.
15. Further observation was conducted 8 weeks after surgery, involving punch biopsies of the anterior vaginal mucosa from three sites. These were then sent on special media to the Anatomical Pathology Laboratory of Dr. M. Djamil General Hospital for examination of the type I/III collagen ratio, MMP-2, and MMP-9.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with second-degree or higher pelvic organ prolapse
2. Postmenopausal pelvic organ prolapse patients
3. Patients with pelvic organ prolapse who will undergo surgery
4. Willingness to participate in the study

Exclusion Criteria:

1. Patients with gynecological malignancies
2. Patients with a history of collagen disease
3. Patients with blood disorders

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Type I/III collagen ratio | From enrollment to the end of treatment at 8 weeks"
  The evaluation of Type I/III collagen ratio are based on imunohistochemistry from punch biopsy in anterior vaginal mucosa that taken durung surgery and at 8 weeks post operative
MMP-2 | From enrollment to the end of treatment at 8 weeks"
  MMP-2 was evaluate based on immunohistochemistry by using punch biopsy of anterior vaginal mucosa during and post surgery
MMP-9 | From enrollment to the end of treatment at 8 weeks"
  MMP-9 are evaluate based on immunohistochemistry from anterior vaginal wall biopsy during and post operative

SECONDARY OUTCOMES:
Pelvic floor muscle strength | From enrollment to the end of treatment at 8 weeks"
  Pelvic floor muscle strength was analyse using biofeedback
Pelvic organ prolapse recurrency | From enrollment to the end of treatment at 8 weeks"
  Pelvic organ prolapse recurrency are evaluate based on POP Q system

CONTACTS AND LOCATIONS:
Overall Officials: Yulia Margaretta Sari Yulia Margaretta, Sari, MD, MD, Principal Investigator — Biomedical Science Doctoral Programme Faculty of Medicine Andalas University/ Urogynecology Division Obstetrics and Gynecology Department M Djamil Hospital Padang Indonesia; Aisyah Elliyanti, Prof, PhD, MD, Study Director — Biomedical Science Doctoral Programme Faculty of Medicine Andalas University; Bobby Indra, Utama, MD, PhD, Study Chair — Biomedical Science Doctoral Programme Faculty of Medicine Andalas University; Zelly Dia, Rofinda, MD, PhD, Study Chair — Biomedical Science Doctoral Programme Faculty of Medicine Andalas University
Locations (1):
- Biomedical Science Doctoral Programme Faculty of Medicine Andalas University/ Urogynecology Division Obstetrics and Gynecology Department M Djamil Hospital Padang, Padang, West Sumatera, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
informed consent should be taken from the patient to share the data

REFERENCES:
- See also: Research protocol — https://bit.ly/45NuVGB
- See also: Research Informed consent — http://bit.ly/45At0qh
- Available data/document: Study Protocol — https://bit.ly/45NuVGB — https://bit.ly/45NuVGB